CLINICAL TRIAL: NCT00117013
Title: A Pilot Trial of Oral Topotecan for the Treatment of Refractory Advanced Solid Neoplasms Expressing HIF-1 Alpha
Brief Title: A Pilot Trial of Oral Topotecan for the Treatment of Refractory Advanced Solid Neoplasms Expressing HIF-1a
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050186; 05-C-0186; NCT00182676 (obsolete NCT alias)
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-08-25

CONDITIONS: Neoplasms
Keywords: Phase I; Antiangiogenesis; Targeted Therapy; Chronic Schedule; VEGF; Cancer; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Topotecan

INTERVENTIONS:
Drug: Fluorine-19-Fluoroded Xyglucose
Drug: Topotecan

SUMMARY:
Background:

HIF-1 is a common mediator of hypoxic and non-hypoxic pathways that affects a transcriptional program leading to survival, angiogenesis, migration and invasion of cancer cells. We have demonstrated that chronic administration of topotecan inhibits HIF-1alpha expression, angiogenesis and tumor growth in human xenografts. Notably, the mechanism by which topotecan inhibits HIF-1alpha protein expression is independent of replication-mediated DNA damage, suggested a mechanism of action distinct from its cytotoxic effects.

Objectives:

This clinical trial is designed to explore the hypothesis that chronic administration of topotecan (TPT) inhibits Hypoxia Inducible factor 1alpha (HIF-1alpha) expression and angiogenesis in patients with metastatic tumors over-expressing HIF-1alpha.

Eligibility:

Adult patients with metastatic solid tumors expressing HIF-1alpha, for whom standard therapy does not exist or would likely not be effective, will be evaluated for study eligibility. Due to safety concerns, pregnant women and HIV-infected individuals are excluded from this study. Prior to enrollment, archival tumor tissue wil be evaluated for the expression of HIF-1alpha as assessed by IHC. Only patients who have tumors that express HIF-1alpha and who meet all eligibility criteria will be enrolled on this study. Patients will be asked to undergo a biopsy to evaluate HIF-1alpha expression before starting treatment and at the end of treatment on cycle 2 (day 12 or 13 cycle 2).

Design:

Topotecan at the dose of 1.2 mg/m(2) will be administered orally daily x 5 for 2 weeks, during a 28 days cycle. Imaging studies including CT, FDG-PET and DCE-MRI will be performed at baseline, at the end of treatment on cycle 1 (day 9 or 10), end of treatment on cycle 2 (day 12 or 13) and then every 2 cycles and will provide information on clinical response as well as tumor metabolism and angiogenesis. The repeat scans on day 9 or 10 of cycle 1 will be performed solely for research purposes to evaluate for early changes in tumor metabolism and angiogenesis. Additional correlative studies include evaluation of mRNA expression of HIF-1 target genes in tumor tissue, circulating markers of angiogenesis, and measurement of circulating endothelial precursor cells (CEP). The goal of this trial is to establish whether topotecan inhibits HIF-1alpha and angiogenesis in human cancers....

DETAILED DESCRIPTION:
Background:

HIF-1 is a common mediator of hypoxic and non-hypoxic pathways that affects a transcriptional program leading to survival, angiogenesis, migration and invasion of cancer cells. We have demonstrated that chronic administration of topotecan inhibits HIF-1alpha expression, angiogenesis and tumor growth in human xenografts. Notably, the mechanism by which topotecan inhibits HIF-1alpha protein expression is independent of replication-mediated DNA damage, suggested a mechanism of action distinct from its cytotoxic effects.

Objectives:

This clinical trial is designed to explore the hypothesis that chronic administration of topotecan (TPT) inhibits Hypoxia Inducible factor 1alpha (HIF-1alpha) expression and angiogenesis in patients with metastatic tumors over-expressing HIF-1alpha.

Eligibility:

Adult patients with metastatic solid tumors expressing HIF-1alpha, for whom standard therapy does not exist or would likely not be effective, will be evaluated for study eligibility. Due to safety concerns, pregnant women and HIV-infected individuals are excluded from this study. Prior to enrollment, archival tumor tissue wil be evaluated for the expression of HIF-1alpha as assessed by IHC. Only patients who have tumors that express HIF-1alpha and who meet all eligibility criteria will be enrolled on this study. Patients will be asked to undergo a biopsy to evaluate HIF-1alpha expression before starting treatment and at the end of treatment on cycle 2 (day 12 or 13 cycle 2).

Design:

Topotecan at the dose of 1.2 mg/m(2) will be administered orally daily x 5 for 2 weeks, during a 28 days cycle. Imaging studies including CT and DCE-MRI will be performed at baseline, at the end of treatment on cycle 1 (day 9 or 10), end of treatment on cycle 2 (day 12 or 13) and will provide information on clinical response as well as tumor angiogenesis. The repeat scans on day 9 or 10 of cycle 1 will be performed solely for research purposes to evaluate for early changes in tumor angiogenesis. Additional correlative studies include evaluation of mRNA expression of HIF-1 target genes in tumor tissue, circulating markers of angiogenesis, and measurement of circulating endothelial precursor cells (CEP). The goal of this trial is to establish whether topotecan inhibits HIF-1alpha and angiogenesis in human cancers.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have a pathologically confirmed solid tumor that is metastatic or unresectable and which has either progressed following standard therapy or for which there is no recommended standard treatment.

Patients must have tumors that can be biopsied with a minimal to small amount of risk and must have a malignancy that expresses HIF-1 alpha protein as measured by immunohistochemistry (determined on archival tissue, at least greater than 10% of cells show positive staining for HIF-1 alpha).

ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).

Life expectancy is greater than 3 months.

Age greater than or equal to 18 years.

Patients must have normal organ and marrow functions as defined below.

* leukocytes greater than or equal to 3000/mm(3).
* absolute neutrophils greater than or equal to 1500/mm(3).
* platelets greater than or equal to 100,000/mm(3).
* AST (SGOT)/ALT (SGPT) less than or equal to 2.5 x institutional upper limit of normal.
* total bilirubin less than or equal to 1.5x institutional upper limit of normal.
* Serum Creatinine less than or equal to 1.5 mg/dL OR creatinine clearance greater than or equal to 50 mL/min for patients with creatinine levels greater than 1.5 mg/dL.
* PT/PTT less than or equal to 1.5 x ULN.

Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.

No unstable medical illness.

Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Patients who have had anticancer therapy (chemotherapy, radiotherapy, vaccines and hormone therapy with the exception of GnRH agonists) within the last 4 weeks (6 weeks for nitrosoureas or mitomycin C or UCN-01); or those who have not recovered from adverse events (reduce to grade 2 or less) due to agents administered more than 4 weeks earlier. Patients must be greater than or equal to 2 weeks since any investigational agent administered as part of a Phase 0 study.

Prior therapy with topotecan.

Patients may not be receiving any other investigational agents. Patients who are on androgen suppression for the treatment of prostate cancer are eligible and will be allowed to continue the androgen suppression therapy on study. No herbal/alternative medications will be allowed on this study other than one multivitamin a day.

Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However, patients who have had treatment for their brain metastases and whose brain metastatic disease has remained stable for at least 4 months without steroids or anti-seizure medications may be enrolled at the discretion of the Principal Investigator.

History of allergic reaction attributed to compounds of similar chemical or biologic composition to topotecan or history of allergic reaction to any component of the topotecan formulation.

Active peptic ulcer or GI condition that could alter absorption or motility.

Pregnant women are excluded from this study. Breastfeeding should be discontinued if the mother is treated with topotecan.

Patients with known immune deficiency syndromes or who are HIV positive will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-06-28; Primary Completion 2010-10-25 (Actual); Study Completion 2010-10-25 (Actual)

PRIMARY OUTCOMES:
To determine whether chronic oral administration of topotecan inhibits HIF-1alpha expression.

SECONDARY OUTCOMES:
To assess tumor angiogenesis in cancers using DCE-MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Semenza GL. Targeting HIF-1 for cancer therapy. Nat Rev Cancer. 2003 Oct;3(10):721-32. doi: 10.1038/nrc1187. PMID 13130303
- [Background] Schioppa T, Uranchimeg B, Saccani A, Biswas SK, Doni A, Rapisarda A, Bernasconi S, Saccani S, Nebuloni M, Vago L, Mantovani A, Melillo G, Sica A. Regulation of the chemokine receptor CXCR4 by hypoxia. J Exp Med. 2003 Nov 3;198(9):1391-402. doi: 10.1084/jem.20030267. PMID 14597738
- [Background] Zhong H, De Marzo AM, Laughner E, Lim M, Hilton DA, Zagzag D, Buechler P, Isaacs WB, Semenza GL, Simons JW. Overexpression of hypoxia-inducible factor 1alpha in common human cancers and their metastases. Cancer Res. 1999 Nov 15;59(22):5830-5. PMID 10582706